CLINICAL TRIAL: NCT04577924
Title: Pre-hospital Care Profile of Road Traffic Injury Victims Presenting to the Emergency Department of a Tertiary Care Centre in Kerala, a Cross-sectional Study
Brief Title: Pre-hospital Care Profile of Road Traffic Injury Victims- Kerala
Acronym: PCP-K
Status: Completed | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Sr. Alphonsa Mathew, Principal Investigator, Jubilee Mission Medical College and Research Institute
Other Study IDs: 36/18/IEC/JMMC&RI; CTRI/2019/03/018160 (Other: Clinical trial registry India)
Record Dates: First submitted 2020-09-29; First posted 2020-10-08 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Trauma; Road (Traffic) Accident [RTA] Nos
MeSH Terms: conditions — Wounds and Injuries | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Road traffic injury victims: All RTI patients presenting to ED within 24 hours of injury is included in the study..
  Individual's not consenting to be part of the study or withdrawing consent later on would be excluded. We also would exclude cases where pre-hospital care provider could not be traced or where reliable data patient could not be collected even after repeated interview.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Trained research assistants would abstract the data as per a preset proforma. The data would be collected from the patient (if coherent), pre-hospital care provider or primary care provider.
  Data would was also obtained from patient records and the proforma filled by the attending doctors on duty.
  Follow up of cases would be done until discharge from the hospital.

SUMMARY:
Selection of appropriate strategies and correct policy-making in these conditions may lead to decreased rates of death due to RTI.There is a lack of research on the effectiveness of pre-hospital care in Kerala. This study aimed to describe the prehospital care of RTI victims presenting to the emergency department in Jubilee Mission Medical College and Research Institute, Thrissur.

DETAILED DESCRIPTION:
Management of trauma is a neglected field in developing nations.Road Traffic Injuries (RTI) cause around 1.35 million deaths worldwide annually according to the statistics of World Health Organization (WHO) and in India 150000 death per year. An overwhelming proportion of these deaths occur before patients even reach the hospital. Two third (60.7%) of the accident victims belonged to the age range of 15 to 44 years. This indicates that active and productive age people are the one affected by road traffic accidents related injuries in turn adding to higher economic loss to the country. Lack of medical attention is attributed to nearly 30 per cent of deaths at site and 80 per cent of the remaining patients died within an hour of injury (golden hour). Most of these deaths are due to airway management failure, respiratory failure or continuing hemorrhage that are preventable causes with appropriate prehospital and subsequent hospital emergency care. Mortality due to RTI is increasing, especially in Low and Middle Income Countries (LMIC). There is a lack of research on the effectiveness of pre-hospital care in India. Selection of appropriate strategies and correct policy-making in these conditions may lead to decreased rates of death due to RTI in several countries.This study aimed to describe the prehospital care of RTI victims presenting to the emergency department (ED) in Jubilee Mission Medical College and Research Institute, Thrissur.

ELIGIBILITY:
Inclusion criteria:

All Road traffic injury (RTI) patients presenting to ED within 24 hours of injury

Exclusion criteria:

Individual's not consenting to be part of the study or withdrawing consent later on

Cases where pre-hospital care provider could not be traced or where reliable patient data could not be collected even after repeated interview.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All RTI patients presenting to ED within 24 hours of injury irrespective of gender, race or comorbidities involved in an RTI would be approached to be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 978 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Pre-hospital care profile of RTI Victims presenting to the emergency department in a tertiary care center in Kerala as measured by a questionnaire. | Hospital admission days through discharge; up to 30 days
  Pre-hospital care received by RTI Victims presenting to the emergency department in a tertiary care center in Kerala

CONTACTS AND LOCATIONS:
Overall Officials: Salish Varghese, MD, Study Chair — salishvarghese@gmail.com
Locations (1):
- Jubilee Mission Medical College and Research Institute, Thrissur, Kerala, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data would be shared once published in a peer reviewed journal.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: from 2025 for a period of 1 year